CLINICAL TRIAL: NCT01724242
Title: Vaginal DHEA to Ease Vaginal Dryness in Women With a Contraindication to Estrogen Therapy
Brief Title: Vaginal DHEA for Women After Breast Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Inability to recruit patients
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DHEA-HMO-CTIL
Record Dates: First submitted 2012-11-07; First posted 2012-11-09 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2015-07

CONDITIONS: Vaginal Dryness; Breast Cancer; Urinary Incontinence; Quality of Life; Sexual Satisfaction
Keywords: Vaginal dryness; Breast Cancer; Urinary Incontinence; Quality of Life; Sexual Satisfaction
MeSH Terms: conditions — Breast Neoplasms; Urinary Incontinence; Orgasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginal DHEA (Experimental): Vaginal DHEA 0.5%(6.5mg)inserted nightly
  Interventions: Drug: Vaginal DHEA
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vaginal DHEA
  Arms: Vaginal DHEA
Drug: Placebo
  Arms: Placebo

SUMMARY:
There does not appear to be a consensus regarding the treatment of vaginal dryness in women who have a contraindication to the use of estrogen products. DHEA, when used locally, may improve the symptoms of vaginal dryness due to its chemical properties.

ELIGIBILITY:
Inclusion Criteria:

* women post menopausal aged 35-55, suffering from vaginal dryness, secondary to chemotherapy for breast cancer, within 5 years of diagnosis. Follicle Stimulating Hormone and Estradiol levels in the post menopausal range are needed.

Exclusion Criteria:

* women using products to alleviate vaginal dryness.
* women taking medication for urinary incontinence
* women not sexually active, for other reasons.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
improvement in vaginal dryness | 12 weeks

SECONDARY OUTCOMES:
improvement in urinary incontinence | 12 weeks
improvement in sexual satisfaction | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Drorith Hochner-Celnikier, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel